CLINICAL TRIAL: NCT01152307
Title: Measuring Quality of Decisions About Treatment of Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Boston (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Carol Cosenza, Project Manager, University of Massachusetts, Boston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CSR-DQ1-002
Record Dates: First submitted 2010-06-22; First posted 2010-06-29 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-07

CONDITIONS: Depression
Keywords: Depression; Depressive disorder; Decision Making; Decision Aids; Decision Quality Instrument
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision Aid (Experimental): Group receiving the decision aid (DVD/booklet)
  Interventions: Behavioral: DVD/Booklet: Coping with Symptoms of Depression
- Control (No Intervention): Group not receiving the decision aid (DVD/booklet)

INTERVENTIONS:
Behavioral: DVD/Booklet: Coping with Symptoms of Depression — DVD and booklet that provides information about treatment choices for depression symptoms
  Other Names: Decision aids; Shared decision making programs
  Arms: Decision Aid

SUMMARY:
The purpose of this randomized controlled trial is to examine the impact of a patient decision aid on the quality of decisions about managing symptoms of depression. In particular, we will examine whether the decision aid increases knowledge about depression/managing depression symptoms and concordance between goals and treatment choices.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+
* In the last 12 months, talked to a health care provider about starting or stopping a treatment (prescription medicine for depression or counseling)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M Gallagher, PhD, Study Director — University of Massachusetts, Boston; Karen R Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Survey Research - University of Massachusetts Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Brodney S, Valentine KD, Sepucha K. Psychometric evaluation of a decision quality instrument for medication decisions for treatment of depression symptoms. BMC Med Inform Decis Mak. 2021 Aug 27;21(1):252. doi: 10.1186/s12911-021-01611-w. PMID 34445969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited through online and newspaper ads by the Center for Survey Research in 17 cities: Atlanta, Baltimore, Boston, Chicago, Dallas-Ft. Worth, Denver, Detroit, Ft. Myers, Houston, Los Angeles, Minneapolis, New York, Phoenix, Portland, Raleigh-Durham, San Francisco, Washington, D.C. August 5, 2010-Jan 10, 2011.
Pre-assignment Details: Eligible patients received a mailed survey and were randomly selected to receive a DVD or no DVD and booklet about depression.
Period: Overall Study
Arm/Group | Decision Aid | Control
Started | 191 | 214
Completed | 191 | 214
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid | Control | Total
Number analyzed (Participants) | 191 | 214 | 405
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 186 | 209 | 395
  >=65 years | 5 | 5 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 39.5 (13.4) | 43.5 (16.8) | 42 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 144 | 266
  Male | 69 | 70 | 139
Region of Enrollment [Number; unit: participants]
  United States | 191 | 214 | 405

OUTCOME MEASURES:

1. Primary Outcome: Depression Knowledge
Description: Total knowledge score from factual questions about depression and methods for managing depression symptoms. Score is the percent of knowledge items answered correctly (0 - 100%).
Time Frame: 2 weeks, on average
Population: Participants were randomized to receive the DVD and booklet.
Measure: Mean (Standard Deviation); unit: percent of correct responses
Arm/Group | Decision Aid | Control
Number analyzed (Participants) | 191 | 214
percent of correct responses | 67.0 (14.1) | 63.6 (12.5)
Statistical Analysis 1: Comparison: Decision Aid vs Control; We tested for a difference in the mean total knowledge score between the decision aid and control groups using independent t-test (2 sided). With 100 patients in each arm, the study had more than 90% power to detect a 10% difference in knowledge assuming a common standard deviation of 18%; Test type: Superiority or Other; p = 0.01, t-test, 2 sided; Mean Difference (Net) = 3.42, 95% CI 2-sided [0.76 to 6.09], Standard Deviation 1.6

2. Secondary Outcome: Value Concordance
Description: Measure of how concordant respondents' actual decisions about treatment for their depression are with their stated beliefs
Time Frame: 2 weeks, on average
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: August 5, 2010 through January 10, 2011.
Arm/Group | Decision Aid | Control
Serious Adverse Events (participants affected / at risk) | 0/191 | 0/214
Other Adverse Events (participants affected / at risk) | 0/191 | 0/214

LIMITATIONS AND CAVEATS:
Those who answered fewer than half of the knowledge questions do not have a total knowledge score (primary outcome).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No